CLINICAL TRIAL: NCT07217197
Title: Wearable Wireless Respiratory Monitoring System That Detects and Predicts Opioid Induced Respiratory Depression
Brief Title: Respiratory Monitoring System That Detects & Predicts OIRD
Acronym: RTM-NIH-SBIR-2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: RTM Vital Signs, LLC (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R44DA059491 (NIH); 4R44DA059491-02 (NIH)
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Respiration Disorders
Keywords: respiratory depression; respiratory monitoring system; tidal volume; minute ventilation; respiratory rate; tracheal sound sensor; opioid induced respiratory depression; breathing
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Post-operative surgical patients routinely managed with opioid medications (Other): This is a non-significant risk clinical trial in 120 patients that are undergoing a surgical procedure that routinely utilizes parenteral and oral opioids for post-operative pain control. We plan to recruit and study a similar number of male/female patients with a range of ages and BMI.
  Interventions: Device: Study to evaluate a Respiratory Monitoring System (RMS) with a Tracheal Sound Sensor (TSS) for detecting and predicting opioid induced respiratory Depression (OIRD).

INTERVENTIONS:
Device: Study to evaluate a Respiratory Monitoring System (RMS) with a Tracheal Sound Sensor (TSS) for detecting and predicting opioid induced respiratory Depression (OIRD). — Expert clinicians will evaluate the ability of the RMS sensor and diagnostic algorithms to detect and predict true OIRD events in post-operative patients routinely managed with opioid medications. Expert clinicians will adjudicate detailed reference data and EMR data to identify a true OIRD event. The definition of a true OIRD event will be based upon the PRODIGY Study definition and RTM definition of a true event. Performance of the RMS will be based upon the sensitivity, specificity, positive predictive value, and negative predictive value for detecting true OIRD events.

SUMMARY:
This study is being conducted to evaluate the ability of the Respiratory Monitoring System (RMS) to detect and predict opioid induced respiratory depression (OIRD) in post-operative surgical patients managed with opioid medications. The ability of the RMS to detect OIRD will be compared to the detection of OIRD using a commercial capnometer, pulse oximeter, airflow monitor, and breathing volume monitor .

We hypothesize the RMS will detect the onset and progression of a true OIRD event with high sensitivity, specificity, positive predictive value, and negative predictive value. A true OIRD event will be determined by the reference device trend data.

RTM Vital Signs, LLC is developing a Respiratory Monitoring System (RMS) that consists of a wearable Trachea Sound Sensor (TSS) and a software application that measures the sounds of air flow within the trachea during inhalation and exhalation and cardiovascular sounds. The sounds of airflow in the trachea are used to continuously monitor a patient's respiratory rate (RR), relative tidal volume (TV), relative minute ventilation (MV), pattern of breathing, duration of apnea in a healthcare setting. The cardiovascular sounds are used to continuously monitor pulse rate and PR variability.

Once commercialized, clinicians will observe the RMS trend data on a smart phone, bedside display, or electronic medical record to determine whether the patient is breathing within their normal range, breathing more than their normal range (hyperventilation), breathing less than their normal range (hypoventilation), or not breathing (apnea). Real-time alerts and alarms will be based upon trends in a patient's rate and depth of breathing, number and duration of apnea events, RTM's Risk-Index-Score, and RTM's machine learning/artificial intelligence methods.

DETAILED DESCRIPTION:
TJU research personnel will be trained by RTM personnel to ensure all questions related to the proper use of the device and study methods are addressed prior to application and use.

Subject Screening:

Patients scheduled for surgery at Thomas Jefferson University Hospital will be screened for recruitment and enrollment. Potential study subjects will be contacted by a research coordinator for pre-screening, screening for inclusion/exclusion criteria, and initial informed consent. The following assessments will be performed as part of the screening and eligibility evaluation:

1. Type of surgery and surgeon that routinely orders opioid medications in the PACU, ICU, intermittent ICU, and general wards of TJUH for post-operative pain control.
2. Review of the subjects' medical history, surgical history, and current medications.
3. Review of the subject's systems to confirm the study subject does not currently have unstable cardiovascular disease, a pulmonary infection, severe asthma, severe bronchitis, or severe emphysema.
4. Demographics (year of birth, gender, and race).
5. Body Mass Index (BMI) calculation (based on subjects' height and weight).

Informed Consent:

Subjects interested in participating in the research study after the initial informed consent discussion will be contacted by a study investigator. An investigator will complete the informal consent process (in-person or virtual). The subject will receive a signed copy of the consent document.

Subject Enrollment:

Subjects will be considered enrolled upon consent. If consent is obtained prior to presenting to TJUH, the subject will be re-evaluated for all inclusion and exclusion criteria. A urine pregnancy test will be performed based upon age and LNMP. If any criteria are not met the subject will be excluded from the study without testing. Any subjects that are withdrawn prior to attaching the RMS and data collection will not count against the total evaluated population.

Data Requirements:

Data regarding demographics, medical/surgical history, current medications, current symptoms, laboratory results, and inclusion / exclusion criteria will be captured prior to commencing study related procedures.

A summary of the study data for analysis is listed below:

1. Subject's age, gender, height, weight, neck circumference, and body mass index (BMI) calculation.
2. Examination of the subject's neck prior to attachment of the TSS onto the skin surface and after removal.
3. Recordings of sounds of airflow in the trachea during inhalation/exhalation and cardiovascular sounds using the RMS.
4. Recordings of Hamilton ventilator pneumotach/capnometer/pulse oximeter measurements of RR, relative TV, relative MV, seconds since last breath (duration of apnea), oxygen saturation, and pulse rate (PR)
5. Recordings of Medtronic Capnostream capnometer/pulse oximeter measurements of RR, carbon-dioxide concentration, pulse rate, hemoglobin oxygen saturation, and seconds since last breath (duration of apnea).
6. Recordings of Senzime ExSpiron 2xi breathing volume monitor measurements of RR, relative TV, and relative MV.

6. Patient data from the TJUH electronic medical record, including date/time/dose of medications delivered, laboratory results, imaging results, medical history, physical examination, diagnostic codes, hospital length of stay, any adverse events, clinical outcomes in the hospital, and clinical outcomes 30 days and 60 days after hospital discharge.

Some study data will be recorded on paper source documents and some data will be recorded on a password protected/encrypted computer and stored in a HIPPA compliant Cloud account.

General Study Procedure Protocol-

Data Collection:

Blinded data will be collected/recorded by research personnel at Thomas Jefferson University Hospital located in center city Philadelphia. RMS breathing data and reference breathing data will be recorded upon admission to the hospital for approximately 15 minutes (baseline), in the PACU for a maximum of 24 hours, and on the general wards, ICU, or intermediate ICU for a maximum of 24 hours.

Baseline Procedure:

Upon admission to the hospital, the TSS's acoustic sensor head (containing two microphones) will be adhered to the study subject's neck above the proximal trachea (midline within the sternal notch or side of the neck) with medical adhesive tape. The sensor's body will be adhered to the skin of the chest wall with medical adhesive tape. RMS data will be transmitted via Bluetooth low energy to a software program on an adjacent tablet computer for recording. RMS data will be recorded with the patient breathing normal RR and TV for approximately 15 minutes. The subject may be asked to breath with a deeper depth of breathing and a more shallow depth of breathing during the baseline recording procedure.

In addition, breathing data will be recorded using a reference volume monitor (ExSpiron 2Xi) and a reference airflow monitor, carbon dioxide monitor, and oxygen saturation monitor (Hamilton C-1 ventilator pneumotach, capnometer, and pulse oximeter). The ExSpiron 2Xi uses an electrical impedance method with electrodes adhered to the chest wall for measuring RR, relative TV and relative MV. The Hamilton uses an airflow sensor, a capnometer, and a pulse oximeter to measure PR, oxygen saturation, RR, apnea duration, and carbon dioxide concentration.

All devices will be removed upon completion of the 15 minute baseline procedure.

Data Collection in the Post-Anesthesia Care Unit (PACU):

TJUH nurses and physicians will manage post-operative surgical patients using routine standard-of-care methods for pain control. Long-acting opioids, short-acting opioids, and non-opioid analgesics will be routinely delivered by PACU nurses to manage a patient's post-operative pain.

Blinded RMS breathing data and time-synced reference breathing data (ExSpiron 2Xi volume data) will be recorded once situated in the PACU. The Medtronic Capnostream's capnometer nasal cannula and pulse oximeter finger probe will also be attached to the patient. Data will be recorded for a maximum of 24 hours while PACU nurses manage the patient's post-operative pain using routine standard-of-care methods.

Data Collection on the General Wards, ICU, or intermediate ICU:

Upon leaving the PACU, RMS breathing data and Medtronic Capnostream breathing data will be recorded on the hospital general wards, ICU, and/or intermediate ICU for a maximum of 24 hours. RMS data will be transmitted via Bluetooth low energy to an adjacent tablet computer for recording.

Time-synced Capnostream capnometer reference data (using a nasal cannula) and pulse oximeter reference data (using a finger probe) will be continuously recorded for a maximum of 24 hours. Time-synced ExSpiron reference data (using electrode pads on chest wall) will be recorded for a maximum of 24 hours.

All research data will be blinded (clinicians will not have access to any research data). TJUH nurses will manage their post-operative surgical patients using routine standard-of-care methods for pain control. Long-acting opioids, short-acting opioids, and non-opioid analgesics will be routinely delivered by ward nurses to manage a patient's post-operative pain.

The TSS, Capnostream nasal cannula, and ExSpiron 2Xi electrode pad set will be removed after a maximum of 24 hours of blinded data collection. The ExSpiron pad set may be removed prior to the 24 hours if requested by the patient.

The TSS will be removed and the skin examined for any evidence of irritation, inflammation, or injury. The area of TSS attachment may be photographed. Recorded RMS data, reference breathing data, and de-identified EMR data will be uploaded to an encrypted HIPPA compliance data base.

Data Analysis:

Recorded Capnostream trend data will be analyzed by experienced clinicians in relationship to medication delivery to identify true OIRD events by 2 methods:. One method of data analysis will use the PRODIGY definition of a true OIRD event: 1) RR less than 5 breaths/minute for greater than 3 minutes, 2) hemoglobin oxygen saturation less than 85% for greater than 3 minutes, 3) a period of apnea lasting greater than 30 seconds, 4) and end-tidal carbon dioxide concentration less than 15 mm Hg or greater than 60 mm Hg, or 5) treatment with naloxone to reverse OIRD. The PRODIGY study observed a 46% incidence of OIRD in hospitalized patients managed with parenteral opioids using the above definition. Another method of data analysis will use RTM's definition of a true OIRD event: 1) RR less than 8 breaths/minute for greater than 3 minutes, 2) hemoglobin oxygen saturation less than 90% for greater than 3 minutes, 3) a period of apnea lasting greater than 15 seconds, 4) an end-tidal carbon dioxide concentration less than 20 mm Hg or greater than 50 mm Hg, or 5) treatment with naloxone to reverse OIRD. Experienced clinicians will adjudicate the RMS data and reference breathing data to identify trend data that is missing, uninterpretable, and/or out-of-range.

The RMS data (RR, relative TV, relative MV, apnea duration, PR) will also be compared/correlated with the Hamilton reference data (RR, TV, MV, apnea duration, PR, carbon dioxide concentration) and the ExSpiron 2Xi reference data (RR, relative TV, relative MV) to determine the accuracy of measurement. The correlation will be determined using mean difference, bias, precision, mean-absolute relative difference, standard deviation, and Bland-Altman plots.

Other Data Collection:

A research coordinator will contact each patient 1 to 3 days after completion of data collection and approximately 30 days and 60 days later to document any adverse events and clinical outcomes. Investigators will review the EPIC electronic medical record in detail to determine time/dose of opioid, sedative, anesthetic, and other medication delivery; and to identify clinical signs/symptoms of clinical deterioration with a focus on OIRD.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical patients routinely managed post-op with opioid medication as their primary analgesic for break through pain.
2. Age ≥ 18 years
3. BMI 20 to 40
4. American Society of Anesthesiologists physical status I, II, and III.
5. Understands written and spoken English language

Exclusion Criteria:

1. Age < 18 years.
2. BMI < 20 or > 40.
3. American Society of Anesthesiologists physical status IV and V.
4. Active Do Not Resuscitate (DNR) order.
5. Does not understand written and spoken English well.
6. Anxiety or claustrophobia related to wearing a face mask or nasal cannula.
7. History of skin irritation or inflammation related to the adhesives or materials used in the TSS sensor, facemask, nasal cannula, or pulse oximeter probe.
8. Active infection or inflammation of the skin above the proximal trachea.
9. Anticipated hospital length of stay less than 24 hours.
10. Excessive facial hair that may prevent attachment of the RMS sensor
11. Unstable cardiovascular or pulmonary function or any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff (e.g., known history of hepatitis B or C).
12. Pregnancy or breast feeding.
13. Current participation in an industry sponsored pharmaceutical study or a medical device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate RMS Trend Data Prior to Each True OIRD Event to Determine the Sensitivity, Specificity, Positive Predictive Value, and Negative Predictive Value for Detecting and Predicting a True OIRD Event. | From placement of the TSS and reference devices to device removal. A maximum of 24 hours of RMS and mask/pneumotach data in the PACU and a maximum of 24 hours of RMS and reference breathing data on the general wards, ICU, or intermediate ICU.
  Evaluate the recorded RMS trend data using a variety of analytical methods (pattern recognition, Risk-Index-Score, machine learning/artificial intelligence) to determine the sensitivity, specificity, positive predictive value, and negative predictive value for detecting a true OIRD event in post-operative surgical patients being managed with opioid medications for pain control.

SECONDARY OUTCOMES:
Correlate RMS breathing data to reference breathing data to determine accuracy and precision of measurement. | Baseline -RMS, Hamilton and ExSpiron reference data (15 min max). PACU- RMS, Hamilton , ExSpiron, and Capnostream reference data (90 min max for mask/pnuemotach). Hospital Wards, ICU, iICU- RMS, ExSpiron and Capnostream (reference data 24 hours max).
  Correlate the RMS breathing data to time-synced Hamilton C-1 ventilator reference data (airflow during inhalation/exhalation, RR, TV, MV, apnea duration, PR, oxygen saturation, carbon dioxide concentration), ExSpiron 2Xi reference data (RR, relative TV, relative MV), and Capnostream reference data (RR, duration of apnea, carbon dioxide concentration, PR, and oxygen saturation) recordings to calculate accuracy and precision.
RMS Safety Endpoint | From TSS adhesion on the neck to removal of the TSS for 26+ hours of wear-time.
  The TSS will be removed from the skin of the neck after 26+ hours of wear-time. A clinician will perform a physical examination of the skin site approximately 10 minutes after removal of the TSS to evaluate for erythema, induration, or any injury of the epidermis or dermis. Research staff will document any allergic reaction, skin irritation, or injury that required premature removal of the TSS or medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marc C Torjman, PhD, Principal Investigator — Thomas Jefferson University; Jeffrey I Joseph, DO, Study Director — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Summary data will be included in peer publications and patent applications. Individual patient data may be included in peer publications but may not be shared with other research scientists until patent applications are submitted and IP secured.

REFERENCES:
- [Background] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Background] Mildh LH, Scheinin H, Kirvela OA. The concentration-effect relationship of the respiratory depressant effects of alfentanil and fentanyl. Anesth Analg. 2001 Oct;93(4):939-46. doi: 10.1097/00000539-200110000-00028. PMID 11574361
- [Background] Yadollahi A, Moussavi ZM. Acoustical respiratory flow. A review of reliable methods for measuring air flow. IEEE Eng Med Biol Mag. 2007 Jan-Feb;26(1):56-61. doi: 10.1109/memb.2007.289122. No abstract available. PMID 17278773